CLINICAL TRIAL: NCT05952778
Title: Reminder Messages for Lung Cancer Screening
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0378; NCI-2023-05185 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2023-07-10; First posted 2023-07-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Skin Flaps; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To test lung cancer screening reminder messages to help adults who 1) 50 to 80 years of age, 2) smoke or have smoked, and 3) do not have history of lung cancer by self-report.

DETAILED DESCRIPTION:
Primary Objectives:

-In this project we will develop, refine, and test reminders for LCS to ensure they are acceptable to patients who have a history of cigarette use.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 40-80 years
* Currently use combustible tobacco products or used combustible tobacco products in the past
* English or Spanish speaker (based on self-report) Or an adult caregiver/care partner or family member of someone with a history of combustible tobacco product use (may participate in focus groups, cognitive interviews, surveys)

Exclusion Criteria:

• History of lung cancer (based on self-report)

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ottawa Acceptability questionnaires | through study completion; an average of 1 year
  Score scale ranges
  Strongly agree Agree Neither agree nor disagree Disagree Strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org